CLINICAL TRIAL: NCT00785213
Title: An Open-Label Drug-Drug Interaction Study to Investigate the Effects of Steady State Quinine on the Single-Dose Pharmacokinetics of Rosiglitazone Maleate in Healthy Volunteers
Brief Title: Drug-Drug Interaction Study Between Quinine Sulfate and Rosiglitazone
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Mutual Pharmaceutical Company, Inc. (Industry)
Collaborators: Cetero Research, San Antonio (Network)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: MPC-001-08-1028; R08-0591
Record Dates: First submitted 2008-10-24; First posted 2008-11-05 (Estimated); Results first posted 2009-11-26 (Estimated); Last update posted 2012-08-07 (Estimated); Status verified 2012-07

CONDITIONS: Healthy
Keywords: rosiglitazone; quinine sulfate; drug interactions; cytochrome p450
MeSH Terms: interventions — Rosiglitazone; Quinine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Rosiglitazone Alone (Active Comparator): Baseline rosiglitazone pharmacokinetics.
  Interventions: Drug: Rosiglitazone 4 mg Tablets
- Rosiglitazone with Steady State Quinine Sulfate (Experimental): Rosiglitazone pharmacokinetics in the presence of steady state quinine sulfate.
  Interventions: Drug: Rosiglitazone 4 mg Tablets; Drug: Quinine Sulfate 324 mg Capsules

INTERVENTIONS:
Drug: Rosiglitazone 4 mg Tablets — Rosiglitazone 4 mg tablet administered as a single oral dose on the morning of Day 1.
  Other Names: Avandia®
  Arms: Rosiglitazone Alone
Drug: Rosiglitazone 4 mg Tablets — Co-administered single oral doses of rosiglitazone 4 mg (1 x 4 mg tablet) and quinine sulfate 648 mg (2 x 324 mg capsules) on the morning of Day 7.
  Other Names: Avandia®
  Arms: Rosiglitazone with Steady State Quinine Sulfate
Drug: Quinine Sulfate 324 mg Capsules — Co-administered single oral doses of rosiglitazone 4 mg (1 x 4 mg tablet) and quinine sulfate 648 mg (2 x 324 mg capsules) on the morning of Day 7.
  Other Names: Qualaquin®
  Arms: Rosiglitazone with Steady State Quinine Sulfate

SUMMARY:
Rosiglitazone is predominantly metabolized by cytochrome P450 (CYP) 2C8. Quinine sulfate is an inhibitor of CYP 2C8. This study will evaluate the effect of multiple doses of quinine sulfate at steady-state on the pharmacokinetics of single-dose rosiglitazone in healthy adult subjects.

DETAILED DESCRIPTION:
Rosiglitazone is predominantly metabolized by cytochrome P450 (CYP) 2C8. Quinine sulfate is an inhibitor of CYP 2C8. This study will evaluate the effect of multiple doses of quinine sulfate at steady-state on the pharmacokinetics of single-dose rosiglitazone in healthy adult subjects.

On study Day 1 after a fast of at least 10 hours, twenty four healthy, non-smoking, non-obese, non-pregnant adult volunteers between the ages of 18 and 45 will be given one oral dose of rosiglitazone (1 x 4 mg tablet). Fasting will continue for 4 hours after the dose. Blood samples will be drawn from all participants before dosing and for 24 hours post-dose at times sufficient to adequately define the pharmacokinetics of rosiglitazone. A 2 day washout period will be completed after the first dose of rosiglitazone on Day 1. On Days 4-7 all subjects will receive a dose of quinine sulfate (2 x 324 mg capsules) every 8 hours starting with the 7:15 a.m. dose on Day 4 and continuing through the 11:15 p.m. dose on Day 7. Doses of quinine sulfate on Days 4-6 will be administered without regard to meals. On the morning of Day 7 after an overnight fast of at least 10 hours, all study participants will receive co-administered doses of rosiglitazone (1 x 4 mg tablet) and quinine sulfate (2 x 324 mg capsules). Fasting will continue for 4 hours after the dose. Blood samples will be drawn from all participants before dosing and for 24 hours post-dose at times sufficient to adequately determine the pharmacokinetics of rosiglitazone. A further goal of this study is to evaluate the safety and tolerability of this regimen in healthy volunteers. Subjects will be monitored throughout participation in the study for adverse reactions to the study drug and/or procedures. Blood pressure (sitting for at least 3 minutes) and pulse will be measured prior to dosing and at 1, 2 and 3 hours after the morning dose of rosiglitazone on Days 1 and 7. Electrocardiograms (EKG) will be recorded on Day 4 before dosing of quinine sulfate and at 1, 2 and 4 hours post-dose and on Day 7 before the co-administered doses of rosiglitazone and quinine sulfate and at 1, 2 and 4 hours post-dose. All adverse events whether elicited by query, spontaneously reported, or observed by clinic staff will be evaluated by the investigator and reported in the subject's case report form.

ELIGIBILITY:
Inclusion Criteria:

* Healthy adults 18-45 years of age
* Non-smoking
* Non-pregnant (post-menopausal, surgically sterile or using effective contraceptive measures)
* Body mass index (BMI) less than or equal to 32
* Medically healthy on the basis of medical history and physical examination
* Hemoglobin > or = to 11.5g/dL
* Completion of the screening process within 28 days prior to dosing
* Provision of voluntary written informed consent

Exclusion Criteria:

* Recent participation (within 28 days) in other research studies
* Recent significant blood donation or plasma donation
* Pregnant or lactating
* Test positive at screening for human immunodeficiency virus (HIV), hepatitis B surface antigen (HbsAg), or hepatitis C virus (HCV)
* Recent (2-year) history or evidence of alcoholism or drug abuse
* History or presence of significant cardiovascular, pulmonary, hepatic, gallbladder or biliary tract, renal, hematologic, gastrointestinal, endocrine, immunologic, dermatologic, neurologic, or psychiatric disease
* Subjects who have used any drugs or substances known to inhibit or induce cytochrome (CYP) P450 enzymes and/or P-glycoprotein (P-gp) within 28 days prior to the first dose and throughout the study
* Drug allergies to quinine sulfate or rosiglitazone

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 23 (Actual)
Dates: Start 2008-09; Primary Completion 2008-10 (Actual); Study Completion 2008-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Matthew Davis, MD, Study Chair — Mutual Pharmaceutical Company, Inc.
Locations (1):
- Cetero Research, East Grand Forks, Minnesota, United States

REFERENCES:
- See also: Recalls, Market Withdrawals and Safety Alerts — http://www.fda.gov/opacom/7alerts.html
- See also: Daily Med - Posting of Recently Submitted Labeling to the FDA — http://dailymed.nlm.nih.gov/dailymed/about.cfm

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Twenty-three (23) healthy, non-smoking, adult male and female volunteers from the community at large were enrolled.
Pre-assignment Details: Thirty-three (33) subjects were screened. Four (4) did not qualify for the study, four (4) did not finish the screening process and two (2) were transferred to another study.
Groups:
- Rosiglitazone Alone, Quinine Alone, Rosiglitazone With Quinine: On the morning of Day 1, subjects received a single dose of rosiglitazone (1 x 4 mg tablet) after an overnight fast of at least 10 hours, followed by a 2 day washout period. On Days 4-7, subjects received a dose of quinine sulfate (2 x 324 mg capsules) every 8 hours beginning at 7:15 am on Day 4 and continuing through the 11:15 p.m. dose on Day 7. On the morning of Day 7, subjects received a single dose of rosiglitazone (1 x 4 mg tablet) along with the morning dose of quinine sulfate ( 2 x 324 mg capsules).
Period: Rosiglitazone Alone
Arm/Group | Rosiglitazone Alone, Quinine Alone, Rosiglitazone With Quinine
Started | 23
Completed | 23
Not Completed | 0
Period: 2 Day Washout Period
Arm/Group | Rosiglitazone Alone, Quinine Alone, Rosiglitazone With Quinine
Started | 23
Completed | 23
Not Completed | 0
Period: Quinine Sulfate Alone
Arm/Group | Rosiglitazone Alone, Quinine Alone, Rosiglitazone With Quinine
Started | 23
Completed | 19
Not Completed | 4
Not completed — Adverse Event | 4
Period: Rosiglitazone With Quinine Sulfate
Arm/Group | Rosiglitazone Alone, Quinine Alone, Rosiglitazone With Quinine
Started | 19
Completed | 18
Not Completed | 1
Not completed — Adverse Event | 1

BASELINE CHARACTERISTICS:
Arm/Group | Rosiglitazone Alone, Quinine Alone, Rosiglitazone With Quinine
Number analyzed (Participants) | 23
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 23
  >=65 years | 0
Age Continuous [Mean (Standard Deviation); unit: years] | 25.61 (7.07)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 9
  Male | 14
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1
  Not Hispanic or Latino | 22
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 1
  White | 20
  More than one race | 0
  Unknown or Not Reported | 1
Region of Enrollment [Number; unit: participants]
  United States | 23

OUTCOME MEASURES:

1. Primary Outcome: Maximum Plasma Concentration (Cmax) of Rosiglitazone
Description: The maximum or peak concentration that rosiglitazone reaches in the plasma.
Time Frame: serial pharmacokinetic blood samples drawn prior to dosing on Days 1 and 7 and then 0.5, 1, 1.5, 2, 2.5, 3, 3.5, 4, 5, 6, 8, 10, 12, 16, 20 and 24 hours after dose administration.
Population: Twenty Three (23) subjects were enrolled in this study. Five (5) subjects withdrew from the study. Pharmacokinetic analyses are based upon data obtained from the eighteen (18) subjects that completed the study.
Measure: Mean (Standard Deviation); unit: ug/mL
Groups:
- Rosiglitazone Alone: On the morning of Day 1, subjects received a single dose of rosiglitazone 4 mg after an overnight fast of at least 10 hours, followed by a 2 day washout period.
- Rosiglitazone With Quinine Sulfate: On the morning of Day 7, subjects received a co-administered single oral dose of rosiglitazone 4 mg and quinine sulfate 648 mg after an overnight fast.
Arm/Group | Rosiglitazone Alone | Rosiglitazone With Quinine Sulfate
Number analyzed (Participants) | 18 | 18
ug/mL | 0.41 (0.08) | 0.43 (0.08)

2. Primary Outcome: Area Under the Concentration Versus Time Curve From Time 0 to Time t [AUC(0-t)]
Description: The area under the plasma concentration versus time curve from time 0 to the time of the last measurable concentration (t), as calculated by the linear trapezoidal rule for rosiglitazone.
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: ug-hr/mL
Arm/Group | Rosiglitazone Alone | Rosiglitazone With Quinine Sulfate
Number analyzed (Participants) | 18 | 18
ug-hr/mL | 1.96 (0.41) | 2.07 (0.45)

3. Primary Outcome: Area Under the Concentration Versus Time Curve From Time 0 Extrapolated to Infinity [AUC(0-∞)]
Description: The area under the plasma concentration versus time curve from time 0 to infinity. [AUC(0-∞)] was calculated as the sum of AUC(0-t) plus the ratio of the last measurable plasma concentration to the elimination rate constant for rosiglitazone.
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: ug-hr/mL
Arm/Group | Rosiglitazone Alone | Rosiglitazone With Quinine Sulfate
Number analyzed (Participants) | 18 | 18
ug-hr/mL | 1.99 (0.43) | 2.10 (0.46)

ADVERSE EVENTS:
Groups:
- Rosiglitazone Alone: On the morning of Day 1, subjects received a single dose of rosiglitazone (1 x 4 mg tablet) after an overnight fast of at least 10 hours, followed by a 2 day washout period.
- Quinine Sulfate Alone: On Days 4-7, subjects received a dose of quinine sulfate 648 mg (2 x 324 mg capsules) every 8 hours beginning with the 7:15 a.m. dose on Day 4 and continuing through the 11:15 p.m. dose on Day 7.
- Rosiglitazone With Quinine Sulfate: On the morning of Day 7, subjects were co-administered a dose of rosiglitazone 4mg and quinine sulfate 648 mg (2 x 324 mg capsules) following an overnight fast of at least 10 hours.
Arm/Group | Rosiglitazone Alone | Quinine Sulfate Alone | Rosiglitazone With Quinine Sulfate
Serious Adverse Events (participants affected / at risk) | 0/23 | 0/23 | 0/19
Other Adverse Events (participants affected / at risk) | 1/23 | 18/23 | 3/19
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Rosiglitazone Alone (N=23) | Quinine Sulfate Alone (N=23) | Rosiglitazone With Quinine Sulfate (N=19)
Cardiac flutter (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0)
Palpitations (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0)
Ear congestion (Ear and labyrinth disorders) | 0 (0) | 1 (1) | 0 (0)
Ear discomfort (Ear and labyrinth disorders) | 0 (0) | 10 (15) | 1 (1)
Hypoacusis (Ear and labyrinth disorders) | 0 (0) | 4 (4) | 0 (0)
Tinnitus (Ear and labyrinth disorders) | 0 (0) | 7 (9) | 0 (0)
Abdominal pain upper (Gastrointestinal disorders) | 0 (0) | 2 (2) | 0 (0)
Diarrhea (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Nausea (Gastrointestinal disorders) | 0 (0) | 5 (6) | 2 (4)
Vomiting (Gastrointestinal disorders) | 0 (0) | 4 (5) | 0 (0)
Chest pain (General disorders) | 0 (0) | 1 (1) | 0 (0)
Fatigue (General disorders) | 0 (0) | 0 (0) | 1 (1)
Feeling hot (General disorders) | 0 (0) | 1 (1) | 1 (1)
Pain (General disorders) | 0 (0) | 1 (1) | 1 (1)
Vessel puncture site pain (General disorders) | 1 (1) | 0 (0) | 0 (0)
Dizziness (Nervous system disorders) | 0 (0) | 7 (9) | 2 (2)
Dysgeusia (Nervous system disorders) | 0 (0) | 3 (3) | 0 (0)
Headache (Nervous system disorders) | 0 (0) | 3 (3) | 2 (2)
Hypoaesthesia (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Tremor (Nervous system disorders) | 0 (0) | 3 (4) | 1 (1)
Paranoia (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1)
Nervousness (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0)
Dysuria (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
Flushing (Vascular disorders) | 0 (0) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days